CLINICAL TRIAL: NCT00713466
Title: The Use of Computer-Assisted Learning Pediatrics Program (CLIPP) in the Pediatric Clerkship
Acronym: CLIPP
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Paola Palma Sisto, Medical College of Wisconsin
Other Study IDs: PRO00006980
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2008-07-31 (Estimated); Status verified 2008-07

CONDITIONS: Learning
Keywords: CLIPP cases; Pediatric clerkship; Standardizing; Students' exposure; Essential; Enhancing; Experience

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: all third year medical students entering their pediatric clerkship at the Medical College of Wisconsin

SUMMARY:
The purpose of this study is to determine if utilizing CLIPP (Computer-Assisted Learning Pediatrics Program) cases in the pediatric clerkship will standardize students' exposure to essential pediatric conditions and enhance their learning experience.

DETAILED DESCRIPTION:
The Computer-Assisted Learning Pediatrics Program was developed by members of the Council on Medical Student Medical Education (COMSEP) and has been very well received by both medical students and faculty. The program is a comprehensive Internet-based learning method designed for use by third year medical students during their pediatric rotation. More than 80 medical schools in the US and Canada have been successfully using the CLIPP cases with an estimated 3000 to 4000 cases being reviewed by students weekly. All third year medical students will be required to complete specific cases, based on gaps identified through review of prior student contact logs. Using the students' own patient contact logs, they will also be strongly encouraged to complete any cases for which they have not met the clerkship requirement. Students will be allowed to complete any other cases they choose. The study proposes that by utilizing CLIPP cases in the pediatric rotation, student exposure to essential pediatric conditions will increase, thereby increasing retention of knowledge and increasing their performance on end of clerkship OSCEs (Observed Structured Clinical Exam) and on NBME Pediatric Subject Exam (shelf exam).

ELIGIBILITY:
Inclusion Criteria:

* all third year medical students will be required to complete a specific number of CLIPP cases as part of their pediatric rotation.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All third year medical students entering their pediatric clerkship at the Medical College of Wisconsin
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
student exposure to essential pediatric conditions will increase, thereby increasing knowledge retention and increasing their performance on end of clerkship exams | 2007-2008 academic year

CONTACTS AND LOCATIONS:
Overall Officials: Paola Palma Sisto, MD, Principal Investigator — Medical College of Wisconsin; Sajani Tipnis, MD, Principal Investigator — Medical College of Wisconsin; Karen Marcdante, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States